CLINICAL TRIAL: NCT07232264
Title: Respiratory and Peripheral Muscle Strength as Predictors of Inhaler Treatment Response in Asthma: A Randomized Comparison of Dry Powder and Metered Dose Inhalers
Brief Title: Respiratory and Peripheral Muscle Strength as Predictors of Inhaler Treatment Response in Asthma: A Comparison of DPI and MDI Devices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bugra Kerget (Other)
Responsible Party: Sponsor-Investigator, Bugra Kerget, Associate Professor of Pulmonary Medicine, Atatürk University Faculty of Medicine, Ataturk University
Organization: Ataturk University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B.30.2ATA.0.01.00/600
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Asthma (Diagnosis)
MeSH Terms: conditions — Asthma; Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MDI Group (Experimental): Participants receive inhaled therapy using metered-dose inhalers (MDIs) containing beclomethasone dipropionate 100 µg + formoterol fumarate 6 µg per actuation, 2 puffs twice daily for one month.
  Interventions: Drug: MDI Inhaler Therapy
- DPI Group (Experimental): Participants receive inhaled therapy using dry powder inhalers (DPIs) (Foster® Nexthaler) containing beclomethasone dipropionate 100 µg + formoterol fumarate 6 µg per inhalation, 2 inhalations twice daily for one month.
  Interventions: Drug: DPI Inhaler Therapy

INTERVENTIONS:
Drug: MDI Inhaler Therapy — Patients in the MDI group received Foster® metered-dose inhaler (MDI) containing beclomethasone dipropionate 100 µg + formoterol fumarate 6 µg per actuation, administered as two puffs twice daily for one month.
  Arms: MDI Group
Drug: DPI Inhaler Therapy — Patients in the DPI group received Foster® Nexthaler dry powder inhaler (DPI) containing beclomethasone dipropionate 100 µg + formoterol fumarate 6 µg per inhalation, administered as two inhalations twice daily for one month.
  Arms: DPI Group

SUMMARY:
Asthma is a chronic respiratory disease characterized by variable airway obstruction. Inhaled therapies are the cornerstone of asthma management, and selecting the appropriate inhaler device is essential for effective treatment. Among available devices, metered dose inhalers (MDIs) and dry powder inhalers (DPIs) are commonly used; however, their effectiveness depends not only on the medication but also on the patient's physiological capacity and inhalation technique.

This prospective randomized study aimed to evaluate the factors influencing inhaler treatment response in newly diagnosed asthma patients. A total of 80 patients with at least a high school education, who demonstrated perfect inhaler technique and adherence, were randomly assigned to MDI or DPI groups (n = 40 each). Baseline and one-month follow-up assessments included pulmonary function tests (PFTs), inspiratory and expiratory muscle strength measurements (MIP, MEP), Asthma Control Test (ACT), and handgrip strength (HGS).

The study investigated how respiratory and peripheral muscle strength, inspiratory capacity, coordination skills, and clinical status affect treatment outcomes with MDI and DPI. Findings from this research may help guide inhaler selection based on patient-specific physiological characteristics to optimize treatment effectiveness.

ELIGIBILITY:
Inclusion Criteria:

Adults aged ≥ 18 years Newly diagnosed asthma according to GINA guidelines Education level of at least high school Ability to use inhaler devices correctly after standardized training Provided written informed consent to participate

Exclusion Criteria:

Presence of other chronic lung diseases (e.g., COPD, interstitial lung disease) Acute asthma exacerbation at the time of enrollment Severe neurological or cognitive impairment affecting inhaler use

Pregnancy or breastfeeding

Refusal or inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-09-24 (Actual); Study Completion 2025-09-24 (Actual)

PRIMARY OUTCOMES:
Change in FEV₁ (%) from Baseline to 1 Month | Baseline and 1 month after treatment initiation
  The primary outcome is the change in forced expiratory volume in one second (FEV₁) expressed as percent of predicted from baseline to one month after initiation of inhaler therapy. Pulmonary function tests were performed according to ATS/ERS 2019 guidelines using the same spirometry device for all participants.

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University, Erzurum, Turkey (Türkiye)